CLINICAL TRIAL: NCT03487536
Title: Nutritional Prognostic Factors in Patients With Amyotrophic Lateral Sclerosis and Percutaneous Endoscopic Gastrostomy
Brief Title: Nutritional Prognostic Factors in ALS
Acronym: PEG-ALS
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Researcher, University of Bari
Other Study IDs: Policlinic Hospital 2, Bari
Record Dates: First submitted 2018-03-19; First posted 2018-04-04 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Nutritional Deficiency; Neuro-Degenerative Disease; Gastrostomy
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutritional assessment — BMI and cholesterol levels evaluation

SUMMARY:
Background. Several nutritional factors have been evaluated as prognostic factors for survival in ALS patients at earlier stages of the disease [body mass index (BMI), body composition expressed as fat free mass (FFM), fat mass (FM), phase angle (PhA), low-density lipoprotein/high-density lipoprotein (LDL/HDL) ratio, cholesterol levels], while only two studies have evaluated some of these parameters after PEG placement.

Aim. BMI and cholesterol levels were evaluated as prognostic factors for survival after percutaneous endoscopic gastrostomy (PEG) placement Moreover, the relationship between body composition and BMI in a subgroup of ALS patients was evaluated.

DETAILED DESCRIPTION:
Methods. Nutritional and neurological parameters were assessed at the time of PEG placement (T0) in 47 consecutive patients. Body composition and PhA were measured in only 22 patients within 2 months from T0. Survival was calculated as the time from the PEG placement to tracheostomy or death.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients who underwent PEG tube placement from 2006 to 2015 and were referred to the artificial nutrition team of the Gastroenterology Unit

Exclusion Criteria:

* ALS patients without PEG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included 47 consecutive patients referring to the Neurological ALS Tertiary Centre, Department of Basic Medical Sciences, Neurosciences and Sense Organs, who underwent PEG tube placement from 2006 to 2015 and were referred to the artificial nutrition team of the Gastroenterology Unit, Department of Emergency and Organ Transplantation, of the same University Hospital. All patients fulfilled revised El Escorial criteria for probable or definite classical ALS.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2006-01-02 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
nutritional assessment | at the time of PEG placement (one day)
  Weight and height (combined to report BMI in kg/m^2)
biochemical nutritional assessment | only at the time of PEG placement (one day)
  cholesterol levels

SECONDARY OUTCOMES:
body composition assessment | within 2 months from the PEG implantation (one day)
  Evaluation of fat mass and fat free mass

CONTACTS AND LOCATIONS:
Overall Officials: Michele Barone, Principal Investigator — University of Bari
Locations (1):
- Policlinic Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided
the results have not yet been shared with all the authors